CLINICAL TRIAL: NCT04269421
Title: Return To Sport Activities in Patients Surgically Treated For Flat Foot in Paeditric Age
Acronym: CSSPORT
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Giovanni Trisolino, MD, Istituto Ortopedico Rizzoli
Other Study IDs: CSSPORT
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Flat Feet; Surgery; Sports Physical Therapy
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: calcaneo-stop: arthrosis of the subtalar joint — arthrosis of the subtalar joint with a screw in the talus bone to stop pathological pronation of the heel
  Other Names: arthrosis of the subtalar joint

SUMMARY:
The SURGERY of arthrosis of the subtalar joint, carried out between 9 and 12 years of age, the aim is to restore and maintain the physiological alignment between the talus and the calcaneus during bone maturation.

There are few articles in the literature that talk about the return to sport of pediatric patients after surgery. The aim of the study is to review patients operated on remotely kick heel and describe how they return in their sports (resilience, type of activities carried out, recovery times). The aim of this study is to evaluate the clinical and functional results of patients of age Pediatric treated in the investigator's SC Orthopedics Pediatric Traumatology department for flat feet with "calcaneostop" surgery. The study aims to describe the method of resuming sports activities, analyzing the timing and difficulties declared by patients after surgery, with the help of specific questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Flatfoot;
* Surgical treatment with arthrorisis of subtalar joint;
* Follow-up> 48 months
* Completeness of the clinical-radiographic documentation.

Exclusion Criteria:

* Diagnosis of secondary flat valgus foot;
* Flat foot treated with other techniques;
* Incomplete clinical documentation;
* Patients who refuse to undergo the study

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The analysis will be performed on pediatric patients undergoing surgical treatment for correction of idiopathic flatfoot in the Orthopedics Pediatric department of the IRCCS Rizzoli Orthopedic Institute in the years 2016-2017.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Patiens Able to Return to Sport After Surgery | 1 year
  timing, sport level, resilience

SECONDARY OUTCOMES:
plantar arch index | 1 year
  The plantar arch index establishes a relationship between the central and posterior regions of the footprint, and it is calculated as follows:A line is drawn tangent to the medial forefoot edge and at the heel region.
  The mean point of this line is calculated. From this mean point, a perpendicular line is drawn crossing the footprint. The same procedure is repeated at the heel tangency. Measurements are obtained of the width of the central region of the footprint (A) and of the heel region (B) in millimeters.
  The plantar arch index is calculated by dividing the A value by B (PAI = A/B).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS - Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided